CLINICAL TRIAL: NCT06272266
Title: Determination of Exercise Capacity and Muscle Strenght in Individuals With COVID-19, the Effect of Aerobic Exercise Training.
Brief Title: The Aerobic Exercise Capacity and Muscle Strenght in Individuals With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selda Sarıkaya (Other)
Collaborators: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Sponsor-Investigator, Selda Sarıkaya, Principal Investigator, Clinical Professor, Bulent Ecevit University
Organization: Bulent Ecevit University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/03-26
Record Dates: First submitted 2022-04-06; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: COVID-19 Pneumonia; COVID-19
Keywords: coronavirus infection; aerobic capacity; cardiopulmonary rehabilitation
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID-19 group (Active Comparator): This group included 32 people aged 18-55 who had previously had COVID-19. Individuals' physical activity levels were measured with the IPAQ short form. Peripheral muscle strength (quadriceps muscle strength, triceps strength, hand grip strength) was measured. The exercise capacities of the individuals were evaluated with a standard exercise tolerance test using a bicycle ergometer. At the end of the test, Borg Scale, test duration, maximum heart rate, maximum work (W) and MET values were recorded. VO2peak levels and VO2peak prediction values were calculated. CPET was applied to 14 people in this group. At the end of the test, the individual's Respiratory Exchange Rate, Anaerobic Threshold, VO2peak, VO2AT (Maximum Oxygen Capacity at Respiratory Anaerobic Threshold), Carbon Dioxide Ventilation Equivalent, heart rate recovery, heart rate recovery in the 1st minute were measured. Aerobic exercise training was given to 14 people in this group. measurements were repeated.
  Interventions: Device: Kardiopulmonary exercise test (Quark KPET C12x/T12x device connected to the Omnia version 1.6.8 COSMED system); Device: Peripheral muscle strength measurement (microFET3 (Hoggan Health Industries, Fabrication Enterprises, lnc) and JAMAR hydraulic hand dynamometer (Sammons Preston, Rolyon, Bolingbrook).; Device: Standard exercise tolerance test (a bicycle ergometer and recorded through the ergoline rehabilitation system 2 Version 1.08 SPI.); Device: Aerobic exercise training (a bicycle ergometer and recorded through the ergoline rehabilitation system 2 Version 1.08 SPI.)
- control group (Active Comparator): This group included 32 people aged 18-55 who had not previously had COVID-19. The physical activity levels of the individuals were measured with the IPAQ short form. Peripheral muscle strength (quadriceps muscle strength, triceps strength, hand grip strength) was measured. The exercise capacities of the individuals were evaluated with a standard exercise tolerance test using a bicycle ergometer. At the end of the test, Borg Scale, test duration, maximum heart rate, maximum work (W) and MET values were recorded. VO2peak levels and VO2peak prediction values were calculated. CPET was applied to 15 people in this group. At the end of the test, the individual's Respiratory Change Rate, Anaerobic Threshold, VO2peak, VO2AT (Maximum Oxygen Capacity at Respiratory Anaerobic Threshold), Carbon Dioxide Ventilation Equivalent, heart rate recovery, Heart rate recovery at 1 minute was measured.
  Interventions: Device: Kardiopulmonary exercise test (Quark KPET C12x/T12x device connected to the Omnia version 1.6.8 COSMED system); Device: Peripheral muscle strength measurement (microFET3 (Hoggan Health Industries, Fabrication Enterprises, lnc) and JAMAR hydraulic hand dynamometer (Sammons Preston, Rolyon, Bolingbrook).; Device: Standard exercise tolerance test (a bicycle ergometer and recorded through the ergoline rehabilitation system 2 Version 1.08 SPI.)

INTERVENTIONS:
Device: Kardiopulmonary exercise test (Quark KPET C12x/T12x device connected to the Omnia version 1.6.8 COSMED system) — For the cardiopulmonary exercise test, a Quark KPET C12x/T12x device connected to the Omnia version 1.6.8 COSMED system, supported by analyzers that measure oxygen uptake and carbon dioxide output, and a bicycle ergometer connected to the ergoline rehab system 2 Version 1.08 SPI system were used. At the end of the test, the individual's RER , VAT, VO2peak, VO2AT, VE/CO2, HRR, HRR1 values were recorded. These values were estimated by the device based on the "wasserman extended" protocol on the Quark KPET C12x/T12x device connected to the Omnia version 1.6.8 COSMED system.The test was repeated after 15 sessions of aerobic exercise training in the Covid-19 group.This intervention was applied to 14 people in the COVID-19 group and 15 people in the control group. It was repeated at the end of 15 sessions of aerobic exercise training in the COVID-19 group.
Device: Peripheral muscle strength measurement (microFET3 (Hoggan Health Industries, Fabrication Enterprises, lnc) and JAMAR hydraulic hand dynamometer (Sammons Preston, Rolyon, Bolingbrook). — Quadriceps and triceps muscle strength was measured in kilograms using the microFET3 (Hoggan Health Industries, Fabrication Enterprises, lnc) manual muscle strength measurement device in the lower and upper extremity. Hand grip strength was evaluated in the dominant upper extremity using a JAMAR hydraulic hand dynamometer (Sammons Preston, Rolyon, Bolingbrook)This intervention was repeated for individuals in both groups at the beginning and at the end of the 15-session aerobic exercise training planned for the COVID-19 group.
Device: Standard exercise tolerance test (a bicycle ergometer and recorded through the ergoline rehabilitation system 2 Version 1.08 SPI.) — At the beginning of this test, resting pulse and blood pressure were measured and recorded. The test was performed following a bicycle ergometer protocol recommended by the American Cardiovascular and Pulmonary Rehabilitation Society. After a 2-minute warm-up period at 0 load (W), a submaximal exercise test was performed by increasing the load by 25 W in 2-minute periods. At the end of the test, exercise intensity was evaluated with the perceived difficulty level (borg scale), test duration, maximum heart rate, maximum work (W). , metabolic equivalent (MET) values were recorded. VO2peak and VO2peakpredictive levels were calculated. This test was repeated for individuals in both groups at the beginning and at the end of the 15-session aerobic exercise training planned for the COVID-19 group.
Device: Aerobic exercise training (a bicycle ergometer and recorded through the ergoline rehabilitation system 2 Version 1.08 SPI.) — Aerobic exercise training was planned for the COVID-19 group with the help of a bicycle ergometer and recorded through the ergoline rehabilitation system 2 Version 1.08 SPI. Aerobic exercise training was applied for a total of 15 sessions, at least 3 days a week, under the supervision of a physician.
  Arms: COVID-19 group

SUMMARY:
The subject of the project is the impact of COVID-19 on the exercise capacity of patients. The long-term sequelae of COVID-19 infection are still unknown. It is not yet clear whether pulmonary sequelae, which may be a consequence of the disease, are associated with a measurable functional deficit. In this project, the aerobic capacity of healthy people will be compared with individuals who have experienced Covid-19, and the amount of increase in aerobic capacity will be determined at the end of 15 sessions by applying a rehabilitation program including bicycle ergometry to individuals who have experienced Covid-19 Detailed description : In December 2020, in the pneumonia epidemic in which the city of Wuhan, China is the center, pneumonia developed due to the newly defined SARS-CoV-2 factor was defined as Coronavirus disease 2019 (COVID-19). It has been observed that clinical findings of SARS-CoV-2 infection in patients hospitalized in Wuhan range from mild manifestations such as asymptomatic disease and mild upper respiratory tract infection to severe viral pneumonia accompanied by respiratory failure and may result in death.The long-term sequelae of COVID19 are still unknown. Pulmonary sequelae that impair physical fitness have been predominantly defined for hospitalized patients with COVID-19. Although lung lesions have been identified as asymptomatically in infected individuals, it is not yet clear whether these observations are related to a measurable functional deficit in physical fitness. They measured the change in the predicted maximum aerobic capacity (VO2 max) of non-infected,asymptomatically infected, and recovering COVID-19 individuals with a well-established and validated physical fitness test before and after the COVID-19 outbreak among young Swiss adults.They demonstrated decreased aerobic capacity in young adults 1 to 2 months after symptomatic COVID-19 without physical strength being affected. In their study, 19% of young adults who recovered after COVID-19 had a VO2 max decrease of more than 10% compared to baseline before infection. It has been identified that decreased VO2 max value is the hallmark of interstitial lung disease. SARS-CoV-2 infection causes lung damage even in asymptomatic cases.

A total of 64 people, including 32 people in 2 groups between the ages of 18-55, who have or have not had corona virus infection, who applied to Bülent Ecevit University Faculty of Medicine Physical Therapy and Rehabilitation or Infectious Diseases outpatient clinics for different reasons, will be included in our project. The research start date is February 2021 and the end date is February 2023. At the beginning of the study, demographic information of the individuals such as gender, age,height, weight, occupation, education, body mass index, physical activity level (international physical activity index-IPAQ), the most used hand (dominant hand) in daily life activities will be recorded. In the control group, resting heart rate, blood pressure, saturation measurement, ECG will be performed before exercise. In addition, in order to evaluate their muscle strength, microFET3 manual muscle measurement device will be used to measure the triceps muscle strength in the upper extremity they actively use, and the quadriceps muscle strength of the same side will be measured, and their grip strength will be measured with the JAMAR hydraulic hand dynamometer. Using the international physical activity index(IPAQ), activity status in daily life will be assessed. The exercise capacity of all individuals will be measured with the aid of the COSMED Quark CPET device using the bicycle ergometry test recommended by the American Society of Cardiovascular and Pulmonary Rehabilitation. In this test, submaximal exercise test will be performed by providing 25 W increase in 2 minutes periods after the warm-up period at 0 load (W) for 2 minutes. In addition, the borg scale obtained at the end of the test, metabolic equivalent of task (MET) and maximum work (W), test duration, maximum heart rate parameters will also be recorded in order to evaluate the exercise capacity.

Individuals who have been confirmed by the previous SARS-COV 2 real-time reverse transcriptase polymerase chain reaction (RT-PCR) test to have coronovirus infection after the test will be included in a treatment program of 15 sessions, at least 3 sessions per week, with bicycle ergometry. After 15 sessions, exercise capacity will be re-evaluated using the cycling test, the aforementioned triceps and grip muscle strengths, V02 max, maximum conjugate (MET), maximum work (w), borg scale, maximum heart rate, test time parameters will be saved again after treatment.

DETAILED DESCRIPTION:
The cardiopulmonary exercise test was also performed on 14 individuals from the control group and 15 individuals in the patient group, and by this test, the respiratory exchange ratio (RER), anaerobic threshold (AT), maximum oxygen capacity (VO 2peak ), maximum ventilatory capacity at anaerobic threshold (VO 2AT ), carbon dioxide ventilatory equivalent (VE/CO 2 ), heart rate recovery (HRR) and heart rate recovery at 1 min (HRR1) parameters were evaluated. The test was repeated after 15 sessions of aerobic exercise training for the individuals in the COVID-19 group who participated in the cardiopulmonary exercise test, and the patients were evaluated using the same parameters.

ELIGIBILITY:
Inclusion Criteria:

* Being a healthy volunteer between the ages of 18-55
* be an independent ambulance

Exclusion Criteria:

* -Not being willing to participate in the study
* Be over 55 years old
* Previous symptomatic or asymptomatic coronavirus infection
* Severe audio-visual loss Unstable cardiovascular, neurological or psychiatric disease
* Pregnancy status
* Active asthma and exacerbation of COPD
* Malignancy Neurodegenerative disease with muscle destruction

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Assessment of Triceps muscle strength by using the Micro FET3 muscle strength device | 3-5 weeks
  Triceps and quadriceps muscle strength; It was measured in kilograms using the microFET3 (Hoggan Health Industries, Fabrication Enterprises, lnc) manual muscle strength measurement device in the dominant upper and lower extremities.
Assessment of Maximum work (watts) ın the standard exercise tolerance test using a bicycle ergometer and recording it via ergoline rehab system 2 Version 1.08 SPI. | 3-5 weeks
  In the standard exercise tolerance test, individuals were subjected to an exercise test by using a bicycle ergometer and recording it via ergoline rehab system 2 Version 1.08 SPI. The maximum work (watts) that the individuals could reach in the standard exercise tolerance test was recorded.The measurement was repeated after 15 sessions of aerobic exercise training in the Covid-19 group.
Assessment of Metabolic Equivalent (MET) in the standard exercise tolerance test using a bicycle ergometer and recording it via ergoline rehab system 2 Version 1.08 SPI. | 3-5 weeks
  In the standard exercise tolerance test, individuals were subjected to an exercise test by using a bicycle ergometer and recording it via ergoline rehab system 2 Version 1.08 SPI. The maximum work (watts) that the individuals could reach in the standard exercise tolerance test was recorded.The measurement was repeated after 15 sessions of aerobic exercise training in the Covid-19 group.
Assessment of VO2peak (ml/kg/min) in the exercise tolerance test using a bicycle ergometer and recording it via ergoline rehab system 2 Version 1.08 SPI. | 3-5 weeks
  In the standard exercise tolerance test, individuals were subjected to exercise testing using a bicycle ergometer and recorded through the ergoline rehabilitation system 2 Version 1.08 SPI. VO2peak was calculated based on the maximum work (watts) that individuals could achieve in the standard exercise tolerance test.The measurement was repeated after 15 sessions of aerobic exercise training in the Covid-19 group
Assessment of VO2peakpredictive (%) in the standard exercise tolerance test using a bicycle ergometer and recording it via ergoline rehab system 2 Version 1.08 SPI. | 3-5 weeks
  In the standard exercise tolerance test, individuals were subjected to exercise testing using a bicycle ergometer and recorded through the ergoline rehabilitation system 2 Version 1.08 SPI. VO2peakpredictive was calculated based on the maximum work (watts) that individuals could achieve in the standard exercise tolerance test.The measurement was repeated after 15 sessions of aerobic exercise training in the Covid-19 group.
Assessment of Hand grip strength (kg) by using a JAMAR hydraulic hand dynamometer (Sammons Preston, Rolyon, Bolingbrook). | 3-5 weeks
  Hand grip strength was evaluated in the dominant upper extremity using a JAMAR hydraulic hand dynamometer (Sammons Preston, Rolyon, Bolingbrook). Two consecutive tests were performed on individuals in a sitting position with shoulders in adduction and neutral rotation, elbows in 90 degrees of flexion, forearm and wrist in 0-30 degrees of extension and 0-15 degrees of ulnar deviation, and the highest grip strength was recorded and evaluated in kilograms.The measurement was repeated after 15 sessions of aerobic exercise training in the Covid-19 group.
Assessment of Exchange Ratio(RER ) by using cardiopulmonary exercise test, a Quark KPET C12x/T12x device connected to the Omnia version 1.6.8 COSMED system, | 3-5 weeks
  For the cardiopulmonary exercise test, a Quark KPET C12x/T12x device connected to the Omnia version 1.6.8 COSMED system, supported by analyzers that measure oxygen uptake and carbon dioxide output, and a bicycle ergometer connected to the ergoline rehab system 2 Version 1.08 SPI system were used. At the end of the test, the individual's RER , VAT, VO2peak, VO2AT, VE/CO2, HRR, HRR1 values were recorded. These values were estimated by the device based on the "wasserman extended" protocol on the Quark KPET C12x/T12x device connected to the Omnia version 1.6.8 COSMED system.The test was repeated after 15 sessions of aerobic exercise training in the Covid-19 group
Assessment of Anaerobik Treshold (VAT) by using cardiopulmonary exercise test with a Quark KPET C12x/T12x device connected to the Omnia version 1.6.8 COSMED system, | 3-5 weeks
  For the cardiopulmonary exercise test, a Quark KPET C12x/T12x device connected to the Omnia version 1.6.8 COSMED system, supported by analyzers that measure oxygen uptake and carbon dioxide output, and a bicycle ergometer connected to the ergoline rehab system 2 Version 1.08 SPI system were used. At the end of the test, the individual's RER , VAT, VO2peak, VO2AT, VE/CO2, HRR, HRR1 values were recorded. These values were estimated by the device based on the "wasserman extended" protocol on the Quark KPET C12x/T12x device connected to the Omnia version 1.6.8 COSMED system.The test was repeated after 15 sessions of aerobic exercise training in the Covid-19 group
Assessment of Maximum Oxygen Capacity (VO2peak) by using cardiopulmonary exercise test with a Quark KPET C12x/T12x device connected to the Omnia version 1.6.8 COSMED system, | 3-5 weeks
  For the cardiopulmonary exercise test, a Quark KPET C12x/T12x device connected to the Omnia version 1.6.8 COSMED system, supported by analyzers that measure oxygen uptake and carbon dioxide output, and a bicycle ergometer connected to the ergoline rehab system 2 Version 1.08 SPI system were used At the end of the test, the individual's RER , VAT, VO2peak, VO2AT, VE/CO2, HRR, HRR1 values were recorded. These values were estimated by the device based on the "wasserman extended" protocol on the Quark KPET C12x/T12x device connected to the Omnia version 1.6.8 COSMED system.The test was repeated after 15 sessions of aerobic exercise training in the Covid-19 group
Assessment of Maximum Oxygen Capacity at Ventilatory Anaerobic Threshold (VO2AT) by using cardiopulmonary exercise test with a Quark KPET C12x/T12x device connected to the Omnia version 1.6.8 COSMED system, | 3-5 weeks
  For the cardiopulmonary exercise test, a Quark KPET C12x/T12x device connected to the Omnia version 1.6.8 COSMED system, supported by analyzers that measure oxygen uptake and carbon dioxide output, and a bicycle ergometer connected to the ergoline rehab system 2 Version 1.08 SPI system were used. At the end of the test, the individual's RER , VAT, VO2peak, VO2AT, VE/CO2, HRR, HRR1 values were recorded. These values were estimated by the device based on the "wasserman extended" protocol on the Quark KPET
Assessment of Carbon Dioxide Ventilatory Equivalent (VE/CO2) by using cardiopulmonary exercise test with a Quark KPET C12x/T12x device connected to the Omnia version 1.6.8 COSMED system, | 3-5 weeks
  For the cardiopulmonary exercise test, a Quark KPET C12x/T12x device connected to the Omnia version 1.6.8 COSMED system, supported by analyzers that measure oxygen uptake and carbon dioxide output, and a bicycle ergometer connected to the ergoline rehab system 2 Version 1.08 SPI system were used. At the end of the test, the individual's RER , VAT, VO2peak, VO2AT, VE/CO2, HRR, HRR1 values were recorded. These values were estimated by the device based on the "wasserman extended" protocol on the Quark KPET
Assessment of Heart Rate Recovery (HRR) by using cardiopulmonary exercise test with a Quark KPET C12x/T12x device connected to the Omnia version 1.6.8 COSMED system, | 3-5 weeks
  For the cardiopulmonary exercise test, a Quark KPET C12x/T12x device connected to the Omnia version 1.6.8 COSMED system, supported by analyzers that measure oxygen uptake and carbon dioxide output, and a bicycle ergometer connected to the ergoline rehab system 2 Version 1.08 SPI system were used. At the end of the test, the individual's RER , VAT, VO2peak, VO2AT, VE/CO2, HRR, HRR1 values were recorded. These values were estimated by the device based on the "wasserman extended" protocol on the Quark KPET
Assessment of Heart Rate Recovery at first minute (HRR1) by using cardiopulmonary exercise test with a Quark KPET C12x/T12x device connected to the Omnia version 1.6.8 COSMED system, | 3-5 weeks
  For the cardiopulmonary exercise test, a Quark KPET C12x/T12x device connected to the Omnia version 1.6.8 COSMED system, supported by analyzers that measure oxygen uptake and carbon dioxide output, and a bicycle ergometer connected to the ergoline rehab system 2 Version 1.08 SPI system were used. At the end of the test, the individual's RER , VAT, VO2peak, VO2AT, VE/CO2, HRR, HRR1 values were recorded. These values were estimated by the device based on the "wasserman extended" protocol on the Quark KPET
Assessment of quadriceps muscle strength by using the Micro FET3 muscle strength device | 3-5 weeks
  Triceps and quadriceps muscle strength; It was measured in kilograms using the microFET3 (Hoggan Health Industries, Fabrication Enterprises, lnc) manual muscle strength measurement device in the dominant upper and lower extremities.

SECONDARY OUTCOMES:
Assessment of Physical activity by using the International Physical Activity Questionnaire (IPAQ) | 3-5 weeks
  International Physical Activity Questionnaire (IPAQ) is a scale based on self-report, developed as a result of research conducted in 12 different countries with the support of WHO (Craig et al., 2003). The short form of the scale consists of 7 items. Through the scale, the time spent by the individual for sitting, walking, and moderate and high intensity physical activities is tried to be determined. The time and day values obtained from the scale are multiplied by the MET value determined for each item and added to the total physical activity time. MET values are calculated as sitting: 1.5 MET, walking: 3.3 MET, moderate physical activity: 4.0 MET, vigorous physical activity: 8.0 MET. With the physical activity value obtained after the calculation, the person is classified according to low, medium or high physical activity level.
Assessment of Test Duration (min) in the standard exercise tolerance test using a bicycle ergometer and recording it via ergoline rehab system 2 Version 1.08 SPI. | 3-5 weeks
  In the standard exercise tolerance test, individuals were subjected to exercise testing using a bicycle ergometer and recorded via the ergoline rehabilitation system 2 Version 1.08 SPI. In the standard exercise tolerance test, the test time completed by individuals was measured and recorded.The measurement was repeated after 15 sessions of aerobic exercise training in the Covid-19 group.
Assessment of Perceived Difficulty by using the Borg Scale | 3-5 weeks
  The Borg scale is a simple numerical list. Participants are asked to rate their exertion on the scale during the exercise test, taking into consideration feelings of physical stress and fatigue, disregarding any factor such as leg pain or breathlessness but focusing on the whole feeling of exertion. This is the original 6 - 20 scale for ratings of perceived exertion.The measurement was repeated after 15 sessions of aerobic exercise training in the Covid-19 group.
Assessment of Maximum heart rate (beats/min) in the standard exercise tolerance test using a bicycle ergometer and recording it via ergoline rehab system 2 Version 1.08 SPI. | 3-5 weeks
  In the standard exercise tolerance test, individuals were subjected to an exercise test by using a bicycle ergometer and recording it via ergoline rehab system 2 Version 1.08 SPI. The maximum heart rate that the individuals could reach in the standard exercise tolerance test was recorded.The measurement was repeated after 15 sessions of aerobic exercise training in the Covid-19 group.
Assessment of Systolic and diastolic blood pressure (mmHg) by using a blood pressure monitor | 3-5 weeks
  Individuals' resting systolic and diastolic blood pressure (mmHg) were measured before and after the exercise test.The measurement was repeated after 15 sessions of aerobic exercise training in the Covid-19 group.
Assessment of resting heart rate (beats/min) by using a a pulse oximeter | 3-5 weeks
  individuals resting heart rate was measured with a pulse oximeter before and after the exercise test.The measurement was repeated after 15 sessions of aerobic exercise training in the Covid-19 group.

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Turkey (Türkiye)